CLINICAL TRIAL: NCT02509455
Title: Quantified Balance Measures During Stance and Gait: Comparison of a New Micro-mechanical Gyro-system (Sensoro Von Hocoma AG) With SwayStar (Balance Int. Innov.) for Measurements of Balance Control of Healthy Controls.
Brief Title: Balance Measures During Stance and Gait: Comparison of Gyroscopic Measurements of Trunk Sway
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-071
Record Dates: First submitted 2015-07-20; First posted 2015-07-28 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: Balance control; Body-mounted sensors; Balance Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal 1: SwayStar device used 1st, Sensoro used 2nd
- Normal 2: Sensoro device used 1st, SwayStar used 2nd

SUMMARY:
To investigate whether an extended version of Valedo®Motion (termed Sensoro for brand management purposes), has the same trunk sway measures similar normal reference values of SwayStar. Offline data analysis of data obtained from Sensoro will be compared to data obtained by SwayStar, a highly accurate and widely accepted system for measuring balance control.

DETAILED DESCRIPTION:
1. Determine a long time recording (over 60s) description of any differences in the drift and noise for the 2 systems during simultaneous recordings with the systems aligned with each other at rest.
2. Compare Sensoro trunk sway measures with those of SwayStar for a battery of 17 stance and gait tasks. The tasks to range from tasks with small velocities (standing on 2 legs eyes open, ca 0.1 deg/s or eyes closed on foam ca.10 deg/s) through tandem and gait tasks with velocities of ca 70 deg/s to the most dynamic with high velocities (rising from a chair, ca 150 deg/sec).
3. Estimate the additional value of adding trunk sway values for the yaw axis as an outcome measure of balance control.
4. Estimate the advantage of adding one or two sensors on the legs to help identify gait balance events and body posture.

ELIGIBILITY:
Inclusion Criteria:

* self reported lack of balance problems (checked by the ability to stand on 1 leg, eyes closed, for at least 14 secs).

Exclusion Criteria:

* orthopaedic problems
* presence of diseases which cause balance problems.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Trunk sway angular velocity and displacement stance and gait tasks. | 1 year
  Is trunk sway angular velocity and displacement measured with SwayStar different when measured with Sensoro for a battery of stance and gait tasks

CONTACTS AND LOCATIONS:
Overall Officials: John HJ Allum, DSc, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Lab for Exp Otoneurology, University Hospital Basel, Basel, Switzerland